CLINICAL TRIAL: NCT01809639
Title: Micronized Oral Progesterone and Effect on Time Symptomatic From Concussion: A Pilot Study
Brief Title: Does Oral Micronized Progesterone Shorten Time of Symptoms From Concussion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Medical Society for Sports Medicine (AMSSM) Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00021983
Record Dates: First submitted 2013-03-07; First posted 2013-03-13 (Estimated); Results first posted 2016-07-14 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Concussion
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Progesterone (Experimental): 400mg of oral micronized progesterone (Prometrium®) on days one, two, and three then 200mg on days four and five
  Interventions: Drug: Progesterone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone
  Other Names: Prometrium
  Arms: Progesterone
Drug: Placebo — Standard placebo
  Arms: Placebo

SUMMARY:
Concussions are a common injury among athletes in the United States. The annual incidence of sports and recreational related traumatic brain injuries in the United States is 1.6 to 3.8 million, and the likelihood of an athlete in a contact sport experiencing a concussion is as high as 20 percent per season. Even mild traumatic brain injury, including concussion, can cause long-term cognitive problems that affect a person's ability to perform daily activities and to return to school or work. Far more concerning is the mounting body of evidence that concussions are not just transient injuries - but have cumulative effects. It has been well established in animal models that progesterone has neuroprotective benefits. Animal studies using progesterone for acute post-injury treatment have demonstrated reduced cerebral edema, reduced neuro-inflammatory markers, decreased neuronal loss, and improved behavioral outcomes. To date, there have been no studies to assess whether or not progesterone will be effective for the treatment of concussions. This double-blind placebo controlled trial will assess the ability of 5 days of oral micronized progesterone (Prometrium®) to shorten the duration of symptoms of an athlete diagnosed with concussion. The investigators hypothesize that athletes treated with progesterone will have faster resolution of their concussive symptoms. The investigators believe this study may be the first clinical trial to show an effective treatment for concussion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a concussion
* A 18 years or older
* Diagnosis < 24 hours from injury
* Consent obtained prior to concussion

Exclusion Criteria:

* Pregnant
* Active breast or reproductive organ cancers
* Allergy to peanuts
* History of or current thrombophlebitis or venous thromboembolic disorder
* Females taking birth control
* Known hypersensitivity or prior adverse reaction to progesterone
* Known liver disease

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Miles, MD, Principal Investigator — Wake Forest University Health Sciences; John A Lucas, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone: 400mg of oral micronized progesterone (Prometrium®) on days one, two, and three then 200mg on days four and five
  Progesterone
- Placebo: Placebo: Standard placebo for 5 days
Period: Overall Study
Arm/Group | Progesterone | Placebo
Started | 18 | 7
Completed | 18 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Placebo | Total
Number analyzed (Participants) | 18 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 7 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 18 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Time (in Days) That a Patient Reports Symptoms From Their Concussion.
Description: The total time that a patient reports symptoms will be assessed. Once the patient reports that they are asymptomatic, the patient will repeat the Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) test to determine if the patient's score has returned to baseline.
Time Frame: From date of injury until date asymptomatic, assessed up to 24 months
Measure: Mean (Standard Error); unit: Days Symptomatic
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 18 | 7
Days Symptomatic | 7.3 (8.64) | 4.5 (1.97)
Statistical Analysis 1: Comparison: Progesterone; Test type: Superiority or Other; p = .42, ANOVA

ADVERSE EVENTS:
Arm/Group | Progesterone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/7
Other Adverse Events (participants affected / at risk) | 0/18 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No